CLINICAL TRIAL: NCT04071223
Title: A Phase II Randomized Trial of Radium-223 Dichloride and Cabozantinib in Patients With Advanced Renal Cell Carcinoma With Bone Metastasis (RadiCal)
Brief Title: Testing the Addition of a New Anti-cancer Drug, Radium-223 Dichloride, to the Usual Treatment (Cabozantinib) for Advanced Renal Cell Cancer That Has Spread to the Bone, RadiCaL Study
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2019-05619; NCI-2019-05619 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); A031801 (Other: Alliance for Clinical Trials in Oncology); A031801 (Other: CTEP); U10CA180821 (NIH)
Record Dates: First submitted 2019-08-26; First posted 2019-08-28 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-12

CONDITIONS: Advanced Renal Cell Carcinoma; Chromophobe Renal Cell Carcinoma; Clear Cell Renal Cell Carcinoma; Collecting Duct Carcinoma; Kidney Medullary Carcinoma; Metastatic Malignant Neoplasm in the Bone; Papillary Renal Cell Carcinoma; Stage IV Renal Cell Cancer AJCC v8; Unclassified Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Specimen Handling; cabozantinib; Magnetic Resonance Spectroscopy; radium Ra 223 dichloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (radium Ra 223 dichloride, cabozantinib s-malate) (Experimental): Patients receive radium Ra 223 dichloride IV over 1 minute on day 1 of cycles 1-6 and cabozantinib S-malate PO QD on days 1-28 of every cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo blood and urine sample collection, bone scan, CT, or MRI, and may undergo FDG-PET or NaF-PET throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Scan; Drug: Cabozantinib S-malate; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Other: Questionnaire Administration; Radiation: Radium Ra 223 Dichloride
- Arm B (cabozantinib s-malate) (Active Comparator): Patients receive cabozantinib S-malate PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo blood and urine sample collection, bone scan, CT, or MRI, and may undergo FDG-PET or NaF-PET throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Scan; Drug: Cabozantinib S-malate; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood and urine sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Scan — Undergo bone scan
  Other Names: Bone Scintigraphy
Drug: Cabozantinib S-malate — Given PO
  Other Names: BMS-907351; Cabometyx; Cometriq; XL 184; XL-184; XL184
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Procedure: Positron Emission Tomography — Undergo FDG-PET or NaF-PET
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Other: Questionnaire Administration — Ancillary studies
Radiation: Radium Ra 223 Dichloride — Given IV
  Other Names: Alpharadin; BAY 88-8223; BAY88-8223; Radium 223 Dichloride; RADIUM RA-223 DICHLORIDE; Radium-223 Chloride; Radium-223 Dichloride; Xofigo
  Arms: Arm A (radium Ra 223 dichloride, cabozantinib s-malate)

SUMMARY:
This phase II trial studies whether adding radium-223 dichloride to the usual treatment, cabozantinib, improves outcomes in patients with renal cell cancer that has spread to the bone. Radioactive drugs such as radium-223 dichloride may directly target radiation to cancer cells and minimize harm to normal cells. Cabozantinib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving radium-223 dichloride and cabozantinib may help lessen the pain and symptoms from renal cell cancer that has spread to the bone, compared to cabozantinib alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the symptomatic skeletal event (SSE)-free survival of metastatic renal cell cancer (mRCC) patients with bone metastases treated with cabozantinib S-malate (cabozantinib) + radium Ra 223 dichloride (radium-223 dichloride) compared to cabozantinib alone.

SECONDARY OBJECTIVES:

I. To investigate the safety, toxicity and tolerability as defined by Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 in patients treated with cabozantinib + radium-223 dichloride compared to cabozantinib alone.

II. To assess SSE-free survival of each treatment arm in predefined sub-groups. III. To assess progression-free survival (PFS) in each treatment arm. IV. To assess overall survival (OS) in each treatment arm. V. To assess time to first SSE (defined as first use of radiation therapy to relieve skeletal symptoms, new symptomatic pathologic vertebral or non-vertebral bone fractures, spinal cord compression, or symptomatic tumor-related orthopaedic surgical intervention) in each treatment arm.

VI. To assess the objective response rate by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.

VII. To assess time to subsequent anti-cancer systemic therapy and type of systemic therapy.

EXPLORATORY QUALITY OF LIFE OBJECTIVES:

I. To compare patient-reported pain as assessed by the Brief Pain Inventory questionnaire (BPI) between patients randomized to cabozantinib versus cabozantinib + radium-223 dichloride at 6 months.

II. To compare patient-reported pain as assessed by the BPI between patients randomized to cabozantinib versus cabozantinib + radium-223 dichloride at other timepoints.

III. To compare overall health-related quality of life as assessed by the Patient-Reported Outcomes Measurement Information Systems (PROMIS) Global Health 10 between patients randomized to cabozantinib versus cabozantinib + radium-223 dichloride.

IV. To compare quality-adjusted survival (overall survival x utility score assessed by European Quality of Life Five Dimension Five Level Scale [EQ5D-5L]) between patients randomized to cabozantinib + radium-223 dichloride.

CORRELATIVE OBJECTIVES:

I. To evaluate changes in the following bone turnover markers between arms:

Ia. Marker of bone formation: P1NP, BSAP. Ib. Marker of bone resorption: CTX, NTX. II. To correlate changes in bone turnover markers with SSE-free survival. III. To assess the immunomodulatory properties of cabozantinib with or without radium-223 dichloride at baseline, during treatment, and at progression.

IV. To identify prognostic and predictive genomic biomarkers of response to cabozantinib and radium-223 dichloride via assessment of tissue, circulating tumor cells (CTCs) and circulating tumor deoxyribonucleic acid (DNA) (cfDNA).

V. To assess the association between bone response according to MD Anderson response criteria and SSE-free survival (FS).

VI. To correlate change in level of total alkaline phosphatase and bone-specific alkaline phosphatase to overall response to cabozantinib + radium-223 dichloride compared to cabozantinib alone.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM A: Patients receive radium Ra 223 dichloride intravenously (IV) over 1 minute on day 1 of cycles 1-6 and cabozantinib S-malate orally (PO) once daily (QD) on days 1-28 of every cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ARM B: Patients receive cabozantinib S-malate PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

All patients undergo blood and urine sample collection, bone scan, computed tomography (CT), or magnetic resonance imaging (MRI), and may undergo fludeoxyglucose (FDG)-positron emission tomography (PET) or sodium fluoride (NaF)-PET throughout the study.

After completion of study treatment, patients are followed up every 6 months for up to 5 years from study registration.

ELIGIBILITY:
Inclusion Criteria:

* Documented histologic or cytologic diagnosis of renal cell cancer (RCC). All subtypes of RCC are eligible including but not limited to clear cell, papillary, chromophobe, translocation, collecting duct carcinoma, medullary carcinoma, and unclassified categories. Enrollment of non-clear cell patients will be limited to 20% of the total sample size (~ 42 patients). Once this goal is met, accrual of non-clear cell patients will be discontinued (a notice will be sent out 2 weeks in advance). Sarcomatoid and rhabdoid differentiation are allowed
* Presence of at least 1 metastatic bone lesion not treated with prior radiation is required.

  * The presence of bone metastases can be detected by computed tomography (CT), magnetic resonance imaging (MRI), Tc-99m bone scan or positron emission tomography (PET) (fludeoxyglucose F-18 [FDG] or sodium fluoride [NaF]) imaging. Patients with non-measurable bone-only disease are allowed. Patients may have received prior radiation therapy for bone metastases or other external radiation >= 7 days prior to registration, as long as they still have at least 1 metastatic bone lesion not treated with radiation. Patients with visceral metastases are allowed, as long as they have at least one untreated bone metastases
* No prior treatment with cabozantinib
* No treatment with any type of small molecular kinase inhibitor (including investigational kinase inhibitors) within 2 weeks or 5 half-lives (whichever is shorter) of registration or receipt of any anti-cancer therapy (including investigational therapy, monoclonal antibodies, cytokine therapy) within 3 weeks of registration
* No prior hemibody external radiotherapy
* No prior therapy with radium-223 dichloride or systemic radiotherapy (such as samarium, strontium)
* No major surgery within 6 weeks of randomization. Procedures such as thoracentesis, paracentesis, percutaneous biopsy, Moh's or other topical skin surgery, Lasik eye surgery are not considered major surgery. Patients who have had a nephrectomy may be registered >= 3 weeks after surgery, providing there are no wound-healing complications. Subjects with clinically relevant ongoing complications from prior surgery are not eligible
* Recovery to baseline or =< grade 1 CTCAE version 5.0 from toxicity related to any prior treatment, unless adverse events are clinically nonsignificant and/or stable on supportive therapy
* The use of osteoclast targeted therapy including either bisphosphonates or denosumab is mandated on this study except in patients with contraindications as determined by the treating investigator, including:

  * Hypocalcemia
  * Hypophosphatemia
  * Renal impairment including those with a glomerular filtration rate (GFR) < 35 mL/min using the Cockcroft-Gault equation or acute renal impairment
  * Hypersensitivity to drug formulation

    * Dental condition or need for dental intervention that per the investigator would increase the risk of osteonecrosis of jaw (ONJ).
    * Use of osteoclast targeted therapy or reason against use needs to be recorded in the electronic case report form (eCRF). Additionally, reason for discontinuation of osteoclast targeted therapy need to be appropriately documented in the eCRF
* Not pregnant and not nursing, because this study involves an investigational agent whose genotoxic, mutagenic and teratogenic effects on the developing fetus and newborn are unknown.

  * Therefore, for women of childbearing potential only, a negative urine pregnancy test done =< 28 days prior to registration is required. A female of childbearing potential is a sexually mature female who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months)
* Age >= 18 years
* Karnofsky performance status >= 60%
* No brain metastases or cranial epidural disease unless adequately treated with radiotherapy, radiosurgery, or surgery and stable for at least 4 weeks prior to registration as documented by MRI or CT imaging or deemed stable by clinical investigator. Treated brain metastases are defined as having no ongoing requirement for steroids and no evidence of progression or hemorrhage after treatment for at least 4 weeks prior to registration as documented by MRI or CT imaging or deemed stable by clinical investigator
* No imminent or established spinal cord compression based on clinical symptoms and/or imaging. In patients with untreated imminent or established spinal cord compression, treatment with standard of care as clinically indicated should be completed at least 2 weeks before registration
* No imminent or impending pathologic fracture based on clinical symptoms and/or imaging. In patients with untreated imminent or impending pathologic fracture, treatment with standard of care as clinically indicated should be completed at least 2 weeks before registration
* No significant, uncontrolled intercurrent or recent illness, including but not limited to the following conditions:

  * Cardiovascular disorders: Symptomatic congestive heart failure, unstable angina pectoris, serious cardiac arrhythmia; uncontrolled hypertension defined as sustained blood pressure > 150 mm Hg systolic or > 100 mm Hg diastolic despite optimal antihypertensive treatment; stroke (including transient ischemic attack), myocardial infarction, or other ischemic event, within 6 months before randomization; thromboembolic event (e.g., deep venous thrombosis, pulmonary embolism) within 1 month before randomization
  * Gastrointestinal disorders: Disorders associated with a high risk of perforation or fistula formation: active inflammatory bowel disease, active diverticulitis, active cholecystitis, active symptomatic cholangitis or active appendicitis, active acute pancreatitis or active acute obstruction of the pancreatic or biliary duct, or active gastric outlet obstruction; abdominal fistula, gastrointestinal perforation, bowel obstruction, or intra-abdominal abscess within 3 months before randomization. Note: Complete healing of an intra-abdominal abscess must be confirmed before randomization
  * No clinically significant hematuria, hematemesis, or hemoptysis, or other history of significant bleeding (e.g., pulmonary hemorrhage) within 3 months before randomization
  * No lesions invading major pulmonary blood vessels
  * No other clinically significant disorders:

    * Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy (with no medications prohibited by this protocol [e.g. drug-drug interactions]) with undetectable viral load within 6 months are eligible for this trial
    * For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy (with no medications prohibited by this protocol [e.g. drug-drug interactions]), if indicated
    * Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load (with no medications prohibited by this protocol [e.g. drug-drug interactions])
    * No serious non-healing wound or ulcer
    * No malabsorption syndrome
    * No uncompensated/symptomatic hypothyroidism
    * No moderate to severe hepatic impairment (Child-Pugh B or C)
    * No requirements for hemodialysis or peritoneal dialysis
    * No history of solid organ transplantation
* No chronic concomitant treatment with strong CYP3A4 inducers or inhibitors. Because the list of these agents is constantly changing, it is important to regularly consult a frequently updated medical reference. Patients may not have received a strong CYP3A4 inducer within 12 days prior to registration nor a strong CYP3A4 inhibitor within 7 days prior to registration
* No concomitant anticoagulation with coumarin agents (e.g., warfarin), direct thrombin inhibitors (e.g., dabigatran), direct factor Xa inhibitor betrixaban, or platelet inhibitors (e.g., clopidogrel). Allowed anticoagulants include:

  * Prophylactic use of low-dose aspirin for cardio-protection (per local applicable guidelines) and low-dose low molecular weight heparins (LMWH).
  * Therapeutic doses of LMWH or anticoagulation with direct factor Xa inhibitors rivaroxaban, edoxaban, or apixaban in subjects without known brain metastases who are on a stable dose of the anticoagulant for at least 1 week before first dose of study treatment without clinically significant hemorrhagic complications from the anticoagulation regimen or the tumor.
* Absolute neutrophil count (ANC) >= 1,500/mm^3
* Platelet count >= 100,000/mm^3
* Hemoglobin >= 9 g/dl (transfusions allowed)
* Calculated (calc.) creatinine clearance >= 30 mL/min using the Cockcroft-Gault equation
* Total bilirubin =< 1.5 x upper limit of normal (ULN), for patients with Gilberts disease =< 3.0 x ULN
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 3.0 x ULN
* Urine protein to creatinine (UPC) ratio =< 2 mg/mg OR 24-hr urine protein < 2 g

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2020-07-29 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Symptomatic skeletal event (SSE)-free survival (FS) | From the date of randomization to the date of the earliest occurrence of SSE or death from any cause, assessed up to 5 years
  SSE-FS distribution will be estimated using the method of Kaplan-Meier by treatment arm. Comparison between the two arms will be performed using a one-sided log-rank test and one-sided p-value less than 0.025 will indicate that the experimental arm is superior to the control arm. SSE-FS will be censored at the date of last SSE assessment for those alive and SSE free. Hazard ratio (experimental over control arm) as well as two-sided 90% confidence interval (CI) for treatment will be estimated using the stratified Cox proportional hazard model with a single treatment covariate.

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 5 years
  Will be determined using Common Terminology Criteria for Adverse Events version 5.0. Adverse events will be summarized and compared between arms using chi-square or fisher exact tests as appropriate.
SSE-FS | From randomization to the date of SSE or death due to any cause, whichever comes first, assessed up to 5 years
  Will be estimated with the Kaplan Meier methodology. Comparison between arms or between predefined groups will be conducted using the log-rank test.
Progression-free survival | From randomization to time of radiographic progression or death due to any cause, whichever occurs first, assessed up to 5 years
  Radiographic progression will be defined by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. Will be estimated with the Kaplan Meier methodology. Comparison between arms or between predefined groups will be conducted using the log-rank test.
Overall survival | From randomization to the date of death due to any cause, assessed up to 5 years
  Will be estimated with the Kaplan Meier methodology. Comparison between arms or between predefined groups will be conducted using the log-rank test. Patients who are alive will be censored at last follow up date.
Time to first SSE | From randomization to the date of first SSE or death due to any cause, assessed up to 5 years
  Will be determined in each treatment. The median estimate to first SSE-FS will be calculated.
Overall response rate (ORR) | Up to 5 years
  Will be defined by RECIST version 1.1. Number and proportion of patients achieving ORR (by RECIST) will be summarized with two-sided 90% CI by treatment arm; comparison between arms will be conducted using chi-square or Fisher's exact test as appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Rana R McKay, Principal Investigator — Alliance for Clinical Trials in Oncology
Locations (47):
- United States (47):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - UC San Diego Moores Cancer Center, La Jolla, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Rush MD Anderson Cancer Center, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - Rush MD Anderson Cancer Center at Rush Oak Park, Oak Park, Illinois
  - University of Chicago Medicine-Orland Park, Orland Park, Illinois
  - UI Health Care Mission Cancer and Blood - Ankeny Clinic, Ankeny, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kansas Cancer Center, Kansas City, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - East Jefferson General Hospital, Metairie, Louisiana
  - LSU Healthcare Network / Metairie Multi-Specialty Clinic, Metairie, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Minnesota Oncology - Burnsville, Burnsville, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - NYP/Weill Cornell Medical Center, New York, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - UPMC-Shadyside Hospital, Pittsburgh, Pennsylvania
  - UT Southwestern Simmons Cancer Center - RedBird, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Fort Worth, Fort Worth, Texas
  - UT Southwestern Clinical Center at Richardson/Plano, Richardson, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm

REFERENCES:
- [Derived] Bade RM, Schehr JL, Emamekhoo H, Gibbs BK, Rodems TS, Mannino MC, Desotelle JA, Heninger E, Stahlfeld CN, Sperger JM, Singh A, Wolfe SK, Niles DJ, Arafat W, Steinharter JA, Jason Abel E, Beebe DJ, Wei XX, McKay RR, Choueri TK, Lang JM. Development and initial clinical testing of a multiplexed circulating tumor cell assay in patients with clear cell renal cell carcinoma. Mol Oncol. 2021 Sep;15(9):2330-2344. doi: 10.1002/1878-0261.12931. Epub 2021 Mar 3. PMID 33604999